CLINICAL TRIAL: NCT00720174
Title: A Phase 1 Study of Doxorubicin and A12 in Advanced Soft Tissue Sarcoma
Brief Title: Cixutumumab and Doxorubicin Hydrochloride in Treating Patients With Unresectable, Locally Advanced, or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00285; NCI-2009-00285 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-16227A; CDR0000600157; 16227A; 16227A (Other: University of Chicago Comprehensive Cancer Center); 8131 (Other: CTEP); N01CM00071 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Adult Angiosarcoma; Adult Desmoplastic Small Round Cell Tumor; Adult Epithelioid Sarcoma; Adult Extraskeletal Myxoid Chondrosarcoma; Adult Extraskeletal Osteosarcoma; Adult Fibrosarcoma; Adult Leiomyosarcoma; Adult Liposarcoma; Adult Malignant Mesenchymoma; Adult Malignant Peripheral Nerve Sheath Tumor; Adult Rhabdomyosarcoma; Adult Synovial Sarcoma; Adult Undifferentiated High Grade Pleomorphic Sarcoma of Bone; Childhood Angiosarcoma; Childhood Desmoplastic Small Round Cell Tumor; Childhood Epithelioid Sarcoma; Childhood Fibrosarcoma; Childhood Leiomyosarcoma; Childhood Liposarcoma; Childhood Malignant Mesenchymoma; Childhood Malignant Peripheral Nerve Sheath Tumor; Childhood Pleomorphic Rhabdomyosarcoma; Childhood Rhabdomyosarcoma With Mixed Embryonal and Alveolar Features; Childhood Synovial Sarcoma; Dermatofibrosarcoma Protuberans; Malignant Adult Hemangiopericytoma; Malignant Childhood Hemangiopericytoma; Metastatic Childhood Soft Tissue Sarcoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma; Untreated Childhood Rhabdomyosarcoma
MeSH Terms: conditions — Hemangiosarcoma; Desmoplastic Small Round Cell Tumor; Sarcoma; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Malignant mesenchymal tumor; Neurofibrosarcoma; Rhabdomyosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Dermatofibrosarcoma; Hemangiopericytoma, Malignant | interventions — cixutumumab; Doxorubicin

ARMS (1):
- Treatment (cixutumumab and doxorubicin hydrochloride) (Experimental): Patients receive cixutumumab IV over 1 hour on days 1, 8, and 15 and doxorubicin hydrochloride IV continuously over 44-52 hours beginning on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may continue to receive cixutumumab in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cixutumumab; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of cixutumumab given together with doxorubicin hydrochloride and to see how well they work in treating patients with unresectable, locally advanced, or metastatic soft tissue sarcoma. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving monoclonal antibody cixutumumab together with doxorubicin hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect safety data about the combination of doxorubicin and Cixitumumab and determine if they can be combined with acceptable toxicity at full doses.

SECONDARY OBJECTIVES:

I. To assess the confirmed response rate (CR + PR as defined by RECIST) of patients with locally advanced or metastatic soft tissue sarcoma when treated with combination doxorubicin and Cixitumumab II. To assess the 3 and 6 month progression free survival rate of patients treated with doxorubicin and Cixitumumab.

III. To assess the progression free survival and overall survival of patients treated with doxorubicin and Cixitumumab.

IV. To evaluate changes in left ventricular ejection fraction assessed by MUGA scan after 2, 4 and 6 cycles of therapy compared to baseline.

OUTLINE: This is a multicenter, dose-escalation study of anti-IGF-1R recombinant monoclonal antibody cixutumumab.

Patients receive cixutumumab intravenously (IV) over 1 hour on days 1, 8, and 15 and doxorubicin hydrochloride IV continuously over 44-52 hours beginning on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may continue to receive cixutumumab in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed soft tissue sarcoma

  * Unresectable disease
  * Locally advanced or metastatic disease
* The following tumor types are not allowed:

  * Embryonal and alveolar rhabdomyosarcoma
  * Gastrointestinal stromal tumor
  * Alveolar soft part sarcoma
  * Clear cell sarcoma
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* No more than 1 prior therapy for sarcoma
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* ANC ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Leukocytes ≥ 3,000/µL
* Total bilirubin ≤ upper limit of normal(ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Fasting serum glucose < 120 mg/dL OR below ULN
* LVEF ≥ 50% by MUGA scan
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after the last dose of anti-IGF-1R recombinant monoclonal antibody IMC-A12
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to anti-IGF-1R recombinant monoclonal antibody IMC-A12
* No poorly controlled diabetes mellitus

  * Patients with a history of diabetes mellitus are eligible provided their blood glucose is within normal range and they are on a stable dietary or therapeutic regimen for this condition
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude compliance with study requirements
* No other concurrent investigational or commercial agents or therapies
* Recovered from all prior therapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior major surgery, hormonal therapy (other than replacement), or hormonal therapy

  * No prior radiotherapy to the heart, mediastinum, or chest wall
* No prior anthracycline therapy or anti-IGF-1R therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) of cixitumumab when administered in a combination regimen with fixed dose doxorubicin hydrochloride, in patients with locally advanced or metastatic soft tissue sarcoma | Up to 2 courses of treatment
  The MTD is defined as the dose of Cixitumumab that induces dose-limiting toxicity (DLT) in no more than 20% of patients.

SECONDARY OUTCOMES:
Changes in cardiac function as measured by MUGA scans of the left ventricular ejection fraction | Baseline to 6 courses of treatment
Confirmed response rate (CR + PR) for comparison with doxorubicin treatment in similar historical patient populations | Up to 6 months
  The mean response probability with 90% credible interval will be reported for those patients treated at the dose of cixitumumab found to be the MTD.
Overall survival | Until death due to any cause, or loss to follow-up, assessed up to 6 months
  Will be estimated using the product-limit method Kaplan and Meier. With point-wise estimates for the 3 and 6-month survival proportions reported with 95% confidence intervals using Greenwood's formula for calculation of the variance.
Progression-free survival | Until documented disease progression or death or loss-to-follow-up, assessed up to 6 months
  Will be estimated using the product-limit method Kaplan and Meier. With point-wise estimates for the 3 and 6-month progression-free survival proportions reported with 95% confidence intervals using Greenwood's formula for calculation of the variance.

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Chugh, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (13):
- United States (13):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Chugh R, Griffith KA, Davis EJ, Thomas DG, Zavala JD, Metko G, Brockstein B, Undevia SD, Stadler WM, Schuetze SM. Doxorubicin plus the IGF-1R antibody cixutumumab in soft tissue sarcoma: a phase I study using the TITE-CRM model. Ann Oncol. 2015 Jul;26(7):1459-64. doi: 10.1093/annonc/mdv171. Epub 2015 Apr 9. PMID 25858498